CLINICAL TRIAL: NCT06230068
Title: ExBRAC - Expressive Writing in Breast Cancer - The Pilot Study
Brief Title: ExBRAC - the Pilot Study
Acronym: ExBRAC-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-07984-01
Record Dates: First submitted 2024-01-08; First posted 2024-01-30 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Quality of Life
Keywords: breast cancer; quality of life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Expressive writing (Other): The intervention consists of expressive writing during 20 minutes. The writing should be of the breast cancer, the treatment or other related topics. The patient is invited to write once every week in a separate place. The intervention ends after four weeks. The written text is not collected.
  Interventions: Other: Expressive writing

INTERVENTIONS:
Other: Expressive writing — See description under arm/group description.

SUMMARY:
The EXBRAC pilot study will investigate the quality of life of patients with breast cancer, and the effect of an intervention with expressive writing. This is a pilot study with two purposes, the first is to create a questionnaire specifically developed for the ExBRAC study, and the second to evaluate the feasibility of the expressive writing.

DETAILED DESCRIPTION:
In the first stage of the study, patients newly diagnosed with breast cancer will be interviewed using a semi-structured method. Based on the transcriptions from the interviews, themes will be gathered and transformed into questions. The questions will be compiled into a questionnaire and an expert group will review the questionnaire to ensure no topic is lacking and an adequate number of response options is present. Lastly, the questionnaire will be face-to-face validated, meaning a patient completes it with a research nurse present to apprehend any ambiguities or questions needing clarification.

In the second part of the pilot study, patients will be included to test the feasibility of the interventions consisting of expressive writing. The intervention consists of expressive writing during 20 minutes. The writing should be of the breast cancer, the treatment or other related topics. The patient is invited to write once every week in a separate place. The intervention ends after four weeks. The written text is not collected. In the pilot study, the intervention will be followed by a telephone call about five weeks after inclusion. To test the feasibility of the intervention, 20 to 25 included patient is considered sufficient.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed breast cancer

Exclusion Criteria:

* Does not understand swedish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-03-26 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Number of included patients that completed the intervention | Five weeks after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Linnea Huss, M.D., Ph. D., Principal Investigator — Region Skane
Locations (1):
- Helsingborg Hospital, Helsingborg, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No